CLINICAL TRIAL: NCT03014830
Title: Effect of Alirocumab on Reverse Cholesterol Transport in Humans
Brief Title: Alirocumab and Reverse Cholesterol Transport
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201612021
Record Dates: First submitted 2016-12-06; First posted 2017-01-09 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Atherosclerosis; Coronary Heart Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Disease | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alirocumab (Active Comparator): Subjects will receive alirocumab for 6 weeks.
  Interventions: Drug: Alirocumab
- Placebos (Placebo Comparator): Subjects will receive placebo for 6 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Alirocumab — 150 mg SQ every 2 weeks
  Other Names: Praluent
  Arms: Alirocumab
Drug: Placebos — Placebo injections SQ every 2 weeks
  Other Names: Placebo
  Arms: Placebos

SUMMARY:
Alirocumab is an injectable treatment for elevated blood cholesterol. The hypothesis of this study is that it also increases cholesterol excretion from the body into the stool, a process sometimes called reverse cholesterol transport. A cholesterol metabolic study will be done before and after 6 weeks of alirocumab treatment. If alirocumab increases reverse cholesterol transport, it is possible that this action provides additional protection from cardiovascular disease.

DETAILED DESCRIPTION:
This study is a single-site, randomized, placebo-controlled clinical trial in which about 24 subjects are expected to complete an 8-week study period. The performance site is Washington University School of Medicine. Even though alirocumab is an approved drug, the investigators consider this to be a phase I trial because it is a physiological study in which the primary endpoint is change in fecal cholesterol excretion and measures of reverse cholesterol transport. It is not a treatment protocol and uses healthy subjects.

Subjects with greater than ideal cholesterol but not taking cholesterol lowering drugs will be studied. All receive whole body cholesterol metabolism tests before and after treatment for 6 weeks with either alirocumab or placebo. Each test takes 2 weeks. On the first day the subjects receive about 35 mg cholesterol-d7 intravenously and blood samples are obtained in order to measure cholesterol turnover rate, pool size, esterification rate, transfer from HDL to LDL and removal from the plasma compartment. Fecal cholesterol excretion and related parameters are measured on days 13 and 14 after a relative steady-state is obtained. During this time the subjects consume a metabolic kitchen diet controlled in cholesterol and phytosterol content and consume oral tracer capsules consisting of cholesterol-d5 and sitostanol-d4. Plasma and stool samples are analyzed by gas chromatography/tandem mass spectrometry to determine daily percent cholesterol excretion from rapidly-mixing body cholesterol pools, fecal cholesterol mass and percent cholesterol absorption. The cholesterol metabolic test is repeated on day 43 and final measurements are made on day 57. Treatment effect, defined as the difference between active and placebo treatments is then calculated. Based on animal data it is expected that alirocumab will increase the efficiency of cholesterol excretion from body pools and the rate of removal of cholesterol ester from plasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or with stable medical or surgical illnesses
* LDL>100 mg/dl.

Exclusion Criteria:

* Triglycerides>250
* Taking drugs affecting lipid metabolism
* Elevated liver function tests
* Diabetes mellitus
* A1c 6.5% or greater
* Pregnant
* Breastfeeding
* Desire for conception in either sex.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in percent cholesterol excretion per day. | Measurements made on days 13-15 (baseline) and days 55-57 (on treatment).
  Percent cholesterol excretion per day is defined as the percent of endogenous rapidly-mixing cholesterol pools excreted per day into the stool.
Change from baseline in removal rate of esterified cholesterol from plasma per day. | Measurements made on days 1-3 (baseline) and days 43-45 (on treatment).
  The removal rate of esterified cholesterol from plasma per day is defined as fractional removal rate of esterified cholesterol from the plasma in pools/day.

SECONDARY OUTCOMES:
Change from baseline in LDL cholesterol | Measurements made on day 15 (baseline) and day 57 (on treatment).
  Reduction in LDL with alirocumab treatment.
Change from baseline in percent cholesterol absorption | Measurements made on days 13-15 (baseline) and days 55-57 (on treatment).
  Percent cholesterol absorption is defined as the percent of intestinal cholesterol absorbed into the body.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Ostlund, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share individual data.